CLINICAL TRIAL: NCT05651399
Title: Comparison in Frequency of Hypotension During Sedation of Propofol and Remimazolam in Spinal Anesthesia in Hip Surgery Patients: a Randomized Controlled Clinical Trial
Brief Title: Comparison in Frequency of Hypotension Between Remimazolam and Propofol in Hip Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hajung Kim, Clinical assistant professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-1713
Record Dates: First submitted 2022-08-12; First posted 2022-12-15 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Remimazolam; Propofol; Orthopedic Procedures; Sedatives; Anesthesia, Spinal
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam (Active Comparator): A maintenance dose of remimazolam is administered for sedation
  Interventions: Drug: Remimazolam
- Propofol (Active Comparator): A maintenance dose of propofol is administered for sedation
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Patients receive remimazolam at a rate of 1 mg/kg/hr. When a patient's MOAA/S reaches 3 or less, the rate of remomazolam is maintained at a rate between 0.3 mg/kr/hr and 1.0 mg/kg/hr until the end of surgery.
  Arms: Remimazolam
Drug: Propofol — Patients are administered propofol with an effect-site concentration of 1.0 mcg/mL to 2.5 mcg/mL by target controlled infusion.
  Arms: Propofol

SUMMARY:
The purpose of this study is to compare the incidence of hypotension between remimazolam and propofol for intraoperative sedation in patients undergoing hip surgery with spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-3
* Patients scheduled for hip joint surgery under spinal anesthesia and sedation with propofol or remimzolam

Exclusion Criteria:

* Patients who refuse to participate in this study
* Patients with uncontrolled high blood pressure, hyperthyroidism, dementia in the inability to communicate, or symptomatic coronary artery disease
* Patients with an allergy to propofol, fentanyl, or bupivacaine
* Patients contraindicated for spinal anesthesia, such as coagulopathy, severe aortic stenosis/mitral stenosis, and active infection on lumbar region
* Patients judged to be inappropriate for this study

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Frequency of hypotension during surgery (1hour) | up to 1 hour after initiation of drug infusion
  mean blood pressure less than 65mmHg

SECONDARY OUTCOMES:
Frequency of hypotension during surgery | Throughout the surgery
  mean blood pressure less than 65mmHg
Total administered phenylephrine | Throughout the surgery
  total dose of phenylephrine administered during surgery
Fluid volume | Throughout the surgery
  Total amount of fluid infused during surgery
Number of hypotensive episodes in the post-anesthesia care unit after surgery | up to 1 hour after postanesthesia care unit entry
  mean blood pressure less than 65mmHg
Complications after surgery | up to 7 days after surgery
  Cardiovascular/neurological/respiratory complications, delirium, impaired renal function, or postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea